CLINICAL TRIAL: NCT06690242
Title: A Multicenter, Randomized,Positive Controlled, and Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of MT1013 Injection in Patients With Chronic Kidney Disease and Secondary Hyperparathyroidism Undergoing Maintenance Hemodialysis
Brief Title: MT1013 Injection for the Treatment of Secondary Hyperparathyroidism in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT1013-II-C03
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Secondary Hyperparathyroidism (SHPT) in Subjects With Chronic Kidney Disease (CKD) on Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MT1013 dose regimen 1 (Experimental): MT1013 injection dose regimen 1 administered intravenously (IV) three times per week for 26 weeks.
  Interventions: Drug: MT1013
- MT1013 dose regimen 2 (Experimental): MT1013 injection dose regimen 2 administered intravenously (IV) three times per week for 26 weeks.
  Interventions: Drug: MT1013
- Etelcalcetide (Active Comparator): Etelcalcetide injection administered intravenously (IV) three times per week for 26 weeks.
  Interventions: Drug: Etelcalcetide Hydrochloride
- Placebo (Placebo Comparator): Placebo administered intravenously (IV) three times per week for 26 weeks;
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT1013 — MT1013 is a novel calcimimetic agent
  Arms: MT1013 dose regimen 1
Drug: MT1013 — MT1013 is a novel calcimimetic agent
  Arms: MT1013 dose regimen 2
Drug: Etelcalcetide Hydrochloride — the already-marketed therapeutic agents
  Arms: Etelcalcetide
Drug: Placebo — The measure does not contain the active ingredients
  Arms: Placebo

SUMMARY:
This is a randomized, positive controlled, and placebo-controlled phase II clinical study to evaluate the efficacy and safety of MT1013 injection in the treatment of chronic kidney disease with secondary hyperparathyroidism (SHPT) undergoing maintenance hemodialysis (MHD) subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject capable of understanding written information ,willing to participate in, and provide a written informed consent;
* 2.Male or female subjects must be at least 18 years old when signing the informed consent;
* 3.The subjects must undergo regular maintenance hemodialysis three times a week for at least three months；
* 4.Dialysate calcium concentration≥1.25 mmol/L (2.5 mEq/L);
* 5.Diagnosed of Secondary Hyperparathyroidism (SHPT), with averaged iPTH ≥400 pg/ml14 days prior to screening;
* 6.Receiving active vitamin D sterols must have had no more than a maximum dose change of 50% within the 1 month prior to screening, remain stable;
* 7.Subject receiving calcium supplements, or phosphate binders must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening, remain stable;

Exclusion Criteria:

* 1.The subjects underwent parathyroidectomy within 6 months prior to screening, or plan to undergo parathyroidectomy or ablation or radiation during the study;
* 2.Gastrointestinal bleeding or peptic ulcer medical history within 6 months prior to screening;
* 3.The body mass index of the subjects was less than 18kg/m2 or greater than 35 kg/m2;
* 4.Subjects with severe uncontrolled hypertension, defined as systolic blood pressure>180 mmHg and/or diastolic blood pressure>110 mmHg(Except for transient blood pressure abnormalities seen during dialysis), despite optimal drug treatment prior to enrollment;
* 5.History of epileptic seizures or ongoing epilepsy related treatment within 1 year prior to screening;
* 6.Subjects with a history of malignant tumors within the past 5 years prior to screening;
* 7.Subjects are allergic or intolerant to any component of the investigational drug or Etelcalcetide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with > 30% reduction from baseline in mean iPTH during the efficacy assessment phase | Weeks 22 to 27, inclusive

SECONDARY OUTCOMES:
Percentage of participants with > 50% reduction from baseline in mean iPTH during the efficacy assessment phase | Weeks 22 to 27, inclusive

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China